CLINICAL TRIAL: NCT00789113
Title: Determination of Bioavailability and Clearance of Lamotrigine-XR by a Stable Isotope Technique
Brief Title: Determination of Absorption and Elimination of Lamotrigine-XR
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0308M51662; IND72642 (Other: FDA)
Record Dates: First submitted 2008-11-07; First posted 2008-11-11 (Estimated); Results first posted 2016-01-20 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2015-12

CONDITIONS: Epilepsy; Seizures; Bipolar Disorder; Bipolar Depression
Keywords: lamotrigine; epilepsy; metabolism; bipolar disorder; bipolar depression; glucuronidation
MeSH Terms: conditions — Epilepsy; Seizures; Bipolar Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Extended Release Lamotrigine (Experimental): Extended Release Lamotrigine
  Interventions: Drug: Extended Release Lamotrigine

INTERVENTIONS:
Drug: Extended Release Lamotrigine

SUMMARY:
People over 65 years of ag break down (metabolize) drugs differently than younger adults. It is not known why this happens or how elderly people absorb or break down these drug differently. These difference may show that elderly individuals need lower doses of medications to avoid possible toxicity. We are interested in studying how yor body absorbs and breaks down your lamotrigine medication. This research may indicate that doses of lamotrigine should be lowered as people get older.

DETAILED DESCRIPTION:
If you agree to be in this study you will be admitted in to the General Clinical Research Center (GCRC) for approximately 24 hours on two different days (Part 1 and Part2). We will need you take a portion of your lamotrigine medication in a special form through a needle in your arm (intravenously). The special form of the drug is the same drug as you normally take except that it has a stable label (a NON-radioactive, naturally occurring atom) on the compound so that we can trace a small amount of the drug through your body. No commercial product of lamotrigine for intravenous use is available because of its poor solubility in water. The intravenous formulation used for this study has a chemical, hydroxypropyl-beta-cyclodextrin, that improves the solubility of lamotrigine in water. This formulation is similar to an intravenous formulation approved for another drug, Sporanox® (itraconazole) that is approved by the FDA. We have obtained approval form the FDA for this intravenous lamotrigine product to be used for research purposes and it has been shown to be safe in more than twenty younger individuals. We will collect fourteen (14) blood samples through a small tube placed into a vein in your arm and collect all of your urine over a period of 24 hours. One blood sample will then be drawn each day for 3 days for a total blood collection of seventeen (17 tubes (totaling approximately 170 mL or 11.5 tablespoons). The samples taken from you will be measured for blood chemistries and concentrations of lmaotrigine and its metabolites resulting from the medication that you take to control your disease (epilepsy or depression)

For the second part of the study, you will be switched from your regular lamotrigine (Lamictal®) to once daily morning dosing of an extended-release formulation of Lamictal-XR® (at the same total daily dose). You will remain on the extended-release lamotrigine (Lamictal-XR) for two weeks, after which you will be re-admitted to the GCRC for 24 hours for Part 2 of the study. Study drug administration and blood and urine sampling will be identical to Part I. The extended-release formulation and your regular lamotrigine have been determined by the manufacturer in preliminary studies to be absorbed the same (bioequivalent0. You will not need to change your total daily dose and will only have to take your lamotrigine once daily with the extended-release product. Your blood levels of lamotrigine will be checked to insure that your are achieving the appropriate concentration with new extended-release product. For this study, you will be given a one-month supply free of charge of the extended-release formulation. After the study is completed, you would return to taking your regular lamotrigine dosing. If the FDA has approved the XR formulation at the end of the study, you and your doctor may decide to keep you on the extended-release form of the drug.

With your consent, a genetics sample, consisting of three (3) additional blood tubes (totaling approximately six teaspoonfuls) will also be collected for a genetic analysis. The genetics sample will be identified with a subject number that corresponds to your other samples. We will use this sample to determine the genetic sequence of DNA that you have that is responsible for encoding proteins that are responsible for breaking down or transporting medications like lamotrigine so that they can be eliminated from your body. You can choose to participate in the main study without taking part in the genetics portion of the study. If you withdraw from the main study, the genetics sample will be discarded with the rest of the samples. if you choose to participate in the genetics portion of the study, we will store the genetics sample indefinitely, however, no testing other than for specific DNA sequences will be done unless we have contact you and received permission to do so.

ELIGIBILITY:
Inclusion Criteria:

* Clinical Diagnosis of Epilepsy or Bipolar Depression
* able to have a venus catheter implanted for blood withdrawal and for intravenous infusion
* equal to or over the age of 65

Exclusion Criteria:

* not on any medication that will interact with lamotrigine e.g. carbamazepine, phenytoin, phenobarbital, valproic acid, St. John's wort, rifampin, tamoxifen

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 12 (Actual)
Dates: Start 2008-11; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rory P Remmel, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Extended Release Lamotrigine
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Extended Release Lamotrigine: Once daily dose of extended release lamotrigine given for two weeks following completion of part I of the study (regular lamotrigine)
Arm/Group | Extended Release Lamotrigine
Number analyzed (Participants) | 12
Age, Customized [Number; unit: participants]
  Age 65 and older | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve (AUC) for Oral Bioavailability of Lamotrigine (LTG
Description: To evaluate the absolute bioavailability of immediate release (IR) and extended release (ER) lamotrigine (LTG) via blood and urine sampling for 24 hour period followed by once a day blood sampling for 3 days following initial dose administration.
Time Frame: 1 week
Measure: Geometric Mean (95% Confidence Interval); unit: µg*h/mL
Groups:
- Immediate Release (IR) Lamotrigine: Study population was on chronic IR lamotrigine therapy and first period of the study was a continuation of standard treatment with IR lamotrigine.
Arm/Group | Immediate Release (IR) Lamotrigine | Extended Release Lamotrigine
Number analyzed (Participants) | 12 | 12
µg*h/mL | 142.8 [92.4 to 220.7] | 132.3 [88.1 to 198.8]

ADVERSE EVENTS:
Arm/Group | Extended Release Lamotrigine
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No